CLINICAL TRIAL: NCT05895305
Title: Prospective Trial of Paclitaxel-Coated Pulmonary Balloon for the Treatment of Benign Airway Obstruction (OXYGEN-1 Trial)
Brief Title: Paclitaxel-Coated Pulmonary Balloon for the Treatment of Benign Airway Stenosis
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Airiver Medical, Inc. (Industry)
Collaborators: Libra Medical (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Oxygen-1
Record Dates: First submitted 2023-05-31; First posted 2023-06-08 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Central Airway Obstruction
Keywords: benign; central airway obstruction; drug coated balloon

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm treated by Airiver Pulmonary DCB (Experimental): subject will be treated by Airiver Pulmonary Drug Coated Balloon (DCB) catheter. The balloon is coated with a paclitaxel drug (3.5ug/mm2).
  Interventions: Combination Product: Paclitaxel-Coated Pulmonary Balloon Catheter

INTERVENTIONS:
Combination Product: Paclitaxel-Coated Pulmonary Balloon Catheter — Subjects with benign airway stenosis will be treated by Airiver pulmonary DCB at index procedure
  Other Names: DCB

SUMMARY:
The goal of this Prospective Trial of Paclitaxel-Coated Pulmonary Balloon for the Treatment of Benign Airway Obstruction (OXYGEN-1) is to evaluate clinical safety and potential efficacy of the Airiver Pulmonary DCB in the treatment of benign central airway stenosis.

DETAILED DESCRIPTION:
Benign central airway stenosis/obstruction, including stenosis of the subglottic area, trachea, and bronchi, is related to significant morbidity due to dyspnea and impaired quality of life. It is hypothesized that Airiver pulmonary drug-coated balloon (DCB) will improve patient outcome in the bronchoscopic treatment of benign airway obstruction, and, as an adjunct to standard of care, will prolong airway patency compared to the standard of care alone. This is a prospective, multi-center, single-arm, open-label, safety & feasibility, OUS first in human study for safety and potential efficacy.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form
2. Stated willingness to comply with all study procedures and availability for the duration of the study
3. Male or female, aged ≥18 old
4. Symptomatic, severe (> 50%) benign CAO (by CT or bronchoscopy)

   1. Stenosis is distal to cricoid and proximal to segmental bronchi
   2. Indicated for balloon dilation only or as an adjunct to standard of care
   3. Includes, but not limited to :

      * Post intubation tracheal stenosis (PITS)
      * Post tracheostomy tracheal stenosis (PTTS)
      * Post lung transplantation stenosis
      * Stenosis related to airway stent
      * Subglottic stenosis (SGS)
      * Stenosis due to tuberculosis

Exclusion Criteria:

1. Malignant CAO
2. Dynamic etiology of benign stenosis such as excessive dynamic airway collapse, tracheobronchomalacia, or stenosis due to external compression
3. Presence of a known perforation at the site of proposed dilation
4. Presence of a known fistula between the tracheobronchial tree and esophagus, mediastinum to pleural space
5. Obstruction not amenable to bronchoscopic dilation in the opinion of the investigator
6. Allergy to paclitaxel or structurally related compounds
7. Severe coagulation disorders or current use of anticoagulant or antiplatelet medication that cannot be safely managed per recommended guidelines prior to the index procedure
8. Acute stricture condition that requires emergent procedure (e.g., immediate dilation)
9. Vasculitis that is not well controlled
10. Inability to tolerate bronchoscopy or contraindication to bronchoscopy, anesthesia, or deep sedation
11. Any anatomical limitation of the head and neck, oral cavity or laryngopharynx that may preclude bronchoscopic evaluation or treatment
12. Patient with active pulmonary infection, including but not limited to: COVID-19, influenza, etc.
13. Any disease or condition that interferes with safe completion of the study, such as severe COPD or severe asthma or pulmonary fibrosis.
14. Patients actively being treated with immunosuppressive therapy or with an active immunosuppressed state due to other treatment or underlying disease.
15. Pregnancy or planning on pregnant during the first 12 months of enrollment in the study
16. Life expectancy <1 year
17. Patient is currently enrolled in other investigational studies. Participation in studies for products approved in the US are not considered investigational

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2023-05-16 (Actual); Primary Completion 2025-10-04 (Actual); Study Completion 2029-10-04 (Estimated)

PRIMARY OUTCOMES:
Primary safety: Freedom from major adverse device events (MADE) post index procedure through 30 days. | 30 days
  MADE is defined as:
  * Airway perforation (Pneumothorax)
  * Pneumomediastinum
  * Massive bleeding
  * Mediastinitis requiring the need for IV antibiotics and / or hospitalization
  * Respiratory distress or asphyxia requiring intubation or reintervention
  * Evidence of negative local tissue reaction to paclitaxel Subjects failing any component of the primary safety endpoint will be considered a safety failure, and subjects who remain event free through 30 days will be considered safety successes. Primary safety will be assessed as the proportion of subjects free from the primary safety event.
Primary efficacy: Freedom from symptom-driven target lesion reintervention (TLR) due to recurrence of stenosis through 6 months | 6 months
  The incidence of subjects free from symptom-driven TLR will be assessed via Kaplan-Meier survival analysis.

SECONDARY OUTCOMES:
Incidence of, and time to, symptom-driven target lesion reintervention through 12 months. | 12 months
  assessed via Kaplan-Meier survival analysis.
Bronchoscopic target lesion patency (Myer-Cotton airway grading system) change through 12 months. | 12 months
  Grade 1 - 0-50% obstruction Grade 2 - 51-70% obstruction Grade 3 - 71-99% obstruction Grade 4 - No detectable lumen.
Spirometry (FEV1) change through 12 months | 12 months
  A spirometry will be compared at baseline vs follow-ups. Lower readings indicate more significant obstruction.
mMRC (Modified Medical Research Council) dyspnea scale change through 12 months | 12 months.
  The grade range is from 0-4. Higher grades indicate worse respiratory disability.
Quality of life (QOL) change: Patient report outcomes (SF-12) through 12 months | 12 months
  Converting SF-12 Item Responses to Physical and Mental Standardized Values. Higher scores indicate better health
Clinical pharmacokinetics of paclitaxel by 10 days | 10 days
  plasma paclitaxel concentration will be assessed per predesignated time points.

CONTACTS AND LOCATIONS:
Overall Officials: Kakha Vacharadze, MD, Principal Investigator — National Center for Tuberculosis and Lung Diseases, Tbilisi State Medical University
Locations (1):
- Israeli-Georgian Medical Research Clinic Helsicore, Tbilisi, Georgia